CLINICAL TRIAL: NCT05237011
Title: Peripartum Anesthetic Management of Patients With Preeclampsia: Prospective Cohort International Observational Study
Brief Title: Peripartum Anesthetic Management of Patients With Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Ioscovich, Director of Obstetric Anesthesia Unit, Shaare Zedek Medical Center
Other Study IDs: 0278-21-SZMC
Record Dates: First submitted 2021-12-30; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Preeclampsia
Keywords: Obstetric Anesthesia; Anesthetic Management; Preeclampsia; Regional Anesthesia; Complication
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will conduct a prospective, observational multicentral international study of perioperative management of patients with preeclampsia. The data will be collected from the maternity files and information systems of the medical centers including obstetric, anesthetic and neonatal parameters according to the attached Excel data table.

Results of the study will help to improve the management of patients with preeclampsia and will help to understand the nature and rate of complications. In addition, the study will help in comparing collected data to the data in the literature and as a result improve the safety of care and service that these patient receive in the institution.

DETAILED DESCRIPTION:
In recent years, there has been a growing interest in anesthetic management of parturients diagnosed with preeclampsia.

The management of patients with preeclampsia is influenced by maternal conditions that include airway changes, coagulation dysfunction and significant hemodynamic changes.

Without changing regular practice the investigators will observe and collect data about: the type of anesthesia during surgery, perioperative monitoring and management of these patients (please see study outcomes). Complications reported in the literature include significant elevated blood pressure during laryngoscopy and development of intracranial hemorrhage, spinal/epidural bleeding during neuraxial anesthesia in patients with preeclampsia, and coagulation abnormalities.

Although the number of patients diagnosed with preeclampsia is estimated at five to ten percent of the general maternity population, there is a lack of prospective studies regarding the anesthetic management, obstetric complications and neonatal outcomes. In most centers the data regarding the rate of general anesthesia for cesarean section, the difficulty in performing neuraxial anesthesia, complications related to coagulation dysfunction and other complications, is limited.

In studies published by gynecologists or neonatologists, there is a significant lack of data relevant to the daily practice of anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* Parturient with diagnosis of preeclampsia for Cesarean Section

Exclusion Criteria:

* No

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parturient with diagnosis of preeclampsia that delivered by cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Type of Anesthesia | Final Type of Anesthesia will be defined during the Cesarean Section (during the operation)
  Final Type of Anesthesia for Cesarean Section including General or Regional Anesthesia

SECONDARY OUTCOMES:
Perioperative anesthetic management | Beginning from preoperative assessment by anesthesiologist to discharge from Post-Anesthesia Care Unit (PACU) / ICU (Intensive Care Unit) assessed up to 5 days
  Different issues of perioperative anesthetic management including aspiration prophylaxis, airway management, induction, maintenance and emergence from anesthesia.
  Perioperative anesthetic management issues including:
  1. Aspiration prophylaxis use: Yes/No; type of medication used.
  2. Airway management: Videolaryngoscopy use: Yes/No; number of attempts.
  3. Induction phase of anesthesia: type of antihypertensive medication, hypnotics, opiates, and neuromuscular blocking agent.
  4. Maintenance phase of anesthesia: type of volatile anesthetics, nitrous oxide or TIVA technique.
  5. Emergence phase of anesthesia: type of neuromuscular reversal agent.
Postoperative pain management | From the start of surgery to the end of postoperative care in recovery unit assessed up to 5 days
  Postoperative pain management according to the visual analog scale (VAS) (0 - no pain to 10 - worst pain)
Invasive monitoring use | During surgery
  Invasive monitoring use during Cesarean Section
Anesthetic complications | Anesthetic complications of patient as result of anesthetic management during the surgery until discharge from the hospital, assessed up to 5 days
  Description of Anesthetic complications
Admission to ICU unit | Admission to during current hospitalization and until discharge from the hospital, assessed up to 5 days
  Admission to Intensive Care Unit (ICU) unit (Yes/No) and duration of admission (days)
Use of blood products | Type and total amount of blood products that administered to patient during the surgery and during the hospitalization, assessed up to 5 days
  Type of blood product administered in perioperative period: RBC - Yes/No; FFP - Yes/No; PLT - Yes/No; CRYO - Yes/No.
  Total amount of each blood product units administered during perioperative period.
Indication for surgery | Indication for Cesarean Section will be defined by obstetrician before the operation
  Indication for Cesarean Section
Obstetric complications | Obstetric complications of patient during the surgery until discharge from the hospital, assessed up to 5 days
  Specific obstetric and maternal complications
Apgar score | Will be defined at 1 and 5 minute after fetal delivery during surgery
  Apgar score at 1 and 5 minutes. Apgar score was published by Virginia Apgar. Measured from 0 to 10. The maximum score is a 10, the lowest score is a 0. Scores a 7 or above is considered in good health, while scores under a 7 may require immediate medical care.
Admission to NICU | Admission to NICU unit during the surgery until maternal discharge from the hospital, assessed up to 5 days
  Number of neonates that required admission to Neonatal Intensive Care Unit (NICU). According to decision of neonatologist that presented during the operation
Neonatal complications | Neonatal complications during the surgery until maternal discharge from the hospital, assessed up to 5 days
  Neonatal complications

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Meedical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui MM, Banayan JM, Hofer JE. Pre-eclampsia through the eyes of the obstetrician and anesthesiologist. Int J Obstet Anesth. 2019 Nov;40:140-148. doi: 10.1016/j.ijoa.2019.04.002. Epub 2019 Apr 13. PMID 31208869
- [Background] Hodgkinson R, Husain FJ, Hayashi RH. Systemic and pulmonary blood pressure during caesarean section in parturients with gestational hypertension. Can Anaesth Soc J. 1980 Jul;27(4):389-94. doi: 10.1007/BF03007461. No abstract available. PMID 7407669
- [Background] Ring L, Landau R, Delgado C. The Current Role of General Anesthesia for Cesarean Delivery. Curr Anesthesiol Rep. 2021;11(1):18-27. doi: 10.1007/s40140-021-00437-6. Epub 2021 Feb 24. PMID 33642943
- [Background] Lee LO, Bateman BT, Kheterpal S, Klumpner TT, Housey M, Aziz MF, Hand KW, MacEachern M, Goodier CG, Bernstein J, Bauer ME; Multicenter Perioperative Outcomes Group Investigators. Risk of Epidural Hematoma after Neuraxial Techniques in Thrombocytopenic Parturients: A Report from the Multicenter Perioperative Outcomes Group. Anesthesiology. 2017 Jun;126(6):1053-1063. doi: 10.1097/ALN.0000000000001630. PMID 28383323
- [Background] Hutcheon JA, Lisonkova S, Joseph KS. Epidemiology of pre-eclampsia and the other hypertensive disorders of pregnancy. Best Pract Res Clin Obstet Gynaecol. 2011 Aug;25(4):391-403. doi: 10.1016/j.bpobgyn.2011.01.006. Epub 2011 Feb 18. PMID 21333604